CLINICAL TRIAL: NCT05238389
Title: Intelligent Robot-mediated Therapy With the MOTORE Device
Brief Title: AI-based Upper Limb Rehabilitation Therapy With MOTORE
Acronym: iMotore
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Irene Giovanna Aprile, Director of the Neurorehabilitation Department, Neurologist, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG-iMotore
Record Dates: First submitted 2022-01-25; First posted 2022-02-14 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic group (Experimental): In the robotic group, patients will undergo a 30-session upper limb robotic rehabilitation using the device MOTORE.
  Interventions: Device: AI-based upper limb robotic therapy

INTERVENTIONS:
Device: AI-based upper limb robotic therapy — Patients will be treated using MOTORE, a robotic device that allows passive, active, and active-assistive planar movements of the shoulder and elbow joints. The intervention will consist of 30 sessions, 1 per day and 5 per week. Therefore, each patient will be treated for 6 weeks
  The parameters of the serious games will be proposed by a Decision Support System (DSS), based on an AI-based algorithm trained using data collected during a previous Randomized Controlled Trial.
  The DSS will be fed, at the enrollment, with patient's demographics, clinical characteristics, clinical scales and kinematic/kinetic data measured by the robot during an evaluation session (unassisted reaching movements) and updated every 2 sessions with kinematic/kinetic data only, to tailor the treatment to the patient's current abilities.
  The therapists will be free to use or not the suggested parameters, on the basis of their previous experience with the robot (over 3 years).
  Other Names: MOTORE

SUMMARY:
Stroke is a common disease with a high disabling impact; it is the world's second leading cause of death and the third leading cause of disability. Robotic therapy has been proposed as a viable approach for the rehabilitation of the upper limb, as a way to increase the amount and the intensity of the therapy, and to standardize the treatment. However, robotic technologies have not yet been used to their full potential in terms of tailoring rehabilitation paths and monitoring the response to treatments. The main goal of the study is to use AI algorithms to (a) predict the recovery of the patients and (b) suggest exercises and parameters to improve the outcomes of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* first ischemic or hemorrhagic stroke (verified by MRI or CT);
* time since stroke onset between 1 and 6 months (subacute phase)
* cognitive abilities adequate to understand the experiments and the follow instructions
* upper limb impairment (Fugl-Meyer Assessment - Upper Extremity score ≤58);

Exclusion Criteria:

* fixed contractions in the affected limb (ankylosis, Modified Ashworth Scale equal to 4);
* inability to understand the instructions required for the study;
* behavioral disorders that may influence therapeutic activity;
* other orthopedic or neurological diseases
* inability or unwillingness to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Agreement between the physiotherapists and the decision support system | Through the study, an average of 10 months
  The number of times a physiotherapist refuses to accept the parameters proposed
System Usability Scale | After a 6-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate usability. It ranges from 0 to 100. Higher scores mean better usability.
Technology Acceptance Model (TAM) | After a 6-week robotic rehabilitation intervention
  It is a self-administered questionnaire to evaluate the acceptance of the provided.
  It comprises several questions rated on a 7-point likert scale.
Likert for Satisfaction | After a 6-week robotic rehabilitation intervention
  Satisfaction will be assessed using a 11-point likert scale. It ranges from 0 to 10. Higher scores mean higher satisfaction.

SECONDARY OUTCOMES:
Changes in Fugl-meyer Assessment Upper Extremity motor functioning | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Changes in Fugl-meyer Assessment Upper Extremity motor functioning | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a stroke-specific, performance-based impairment index. It ranges from 0 (hemiplegia) to 66 points (normal).
Changes in Box and Block test (BBT) | Before the intervention, after a 3-week robotic rehabilitation intervention
  The BBT is a standard measure for evaluating manual dexterity. The participants grasp and transfer one-inch square blocks from one compartment to the other, transferring as many as possible. The number of blocks transferred from one side to the other within 1 min is recorded.
Changes in Box and Block test (BBT) | Before the intervention, after a 6-week robotic rehabilitation intervention
  The BBT is a standard measure for evaluating manual dexterity. The participants grasp and transfer one-inch square blocks from one compartment to the other, transferring as many as possible. The number of blocks transferred from one side to the other within 1 min is recorded.
Changes in Action Research Arm Test (ARAT) | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a valid measure of upper-extremity functional limitation. The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance.
Changes in Action Research Arm Test (ARAT) | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a valid measure of upper-extremity functional limitation. The total score on the ARAT ranges from 0 to 57, with the lowest score indicating that no movements can be performed, and the upper score indicating normal performance.
Change in Medical Research Council (MRC) | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a validated measure of strength clinically measured. It ranges from 0, paralysis, to 5, normal strength.
Change in Medical Research Council (MRC) | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of strength clinically measured. It ranges from 0, paralysis, to 5, normal strength.
Change in Frenchay Arm Test | Before the intervention, after a 3-week robotic rehabilitation intervention
  The Frenchay Arm Test (FAT) is a measure of upper extremity proximal motor control and dexterity during activities of daily living in patients with upper limb impairments. The total scores range from 0 to 5 (normal performance).
Change in Frenchay Arm Test | Before the intervention, after a 6-week robotic rehabilitation intervention
  The Frenchay Arm Test (FAT) is a measure of upper extremity proximal motor control and dexterity during activities of daily living in patients with upper limb impairments. The total scores range from 0 to 5 (normal performance).
Change in Modified Ashworth Scale | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a validated measure of spasticity. It ranges from 0 (normal) to 4 (rigid limb).
Change in Modified Ashworth Scale | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of spasticity. It ranges from 0 (normal) to 4 (rigid limb).
Changes in Motricity Index for upper extremity | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a validated measure of upper limb strength. It ranges from 0 (worse) to 100 (normal strength).
Changes in Motricity Index for upper extremity | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated measure of upper limb strength. It ranges from 0 (worse) to 100 (normal strength).
Changes in Numeric Rating Scale for pain | Before the intervention, after a 3-week robotic rehabilitation intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Changes in Numeric Rating Scale for pain | Before the intervention, after a 6-week robotic rehabilitation intervention
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale, from 0 (no pain) to 10 (worst pain imaginable).
Changes in Neuropathic Pain 4 Questions (DN4) | Before the intervention, after a 3-week robotic rehabilitation intervention
  It is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Changes in Neuropathic Pain 4 Questions (DN4) | Before the intervention, after a 6-week robotic rehabilitation intervention
  It is a validated clinician-administered screening tool for neuropathic pain. It ranges from 0 to 10; higher values means higher neuropathic pain probability.
Changes in Modified Barthel Index | Before the intervention, after a 3-week robotic rehabilitation intervention
  The modified is an ordinal scale used to measure performance in activities of daily living. It ranges from 0 to 100, with lower scores indicating increased disability.
Changes in Modified Barthel Index | Before the intervention, after a 6-week robotic rehabilitation intervention
  The modified is an ordinal scale used to measure performance in activities of daily living. It ranges from 0 to 100, with lower scores indicating increased disability.
Changes in 36-Item Short Form Survey (SF-36) | Before the intervention, after a 6-week robotic rehabilitation intervention
  The 36-Item Short Form Survey (SF-36) is a self-reported measure of health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The scores are: vitality; physical functioning; bodily pain; general health perceptions; physical role functioning; emotional role functioning; social role functioning; mental health.
  Moreover, two composite scores, i.e., the Physical Composite Score and the Mental Composite Score, both ranging from 0 to 100, will be considered.
Changes in the Duration Index. | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Duration" is the time required to complete the task. It is measured in seconds.
Changes in the Duration Index. | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Duration" is the time required to complete the task. It is measured in seconds.
Changes in Velocity_mean Index. | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Velocity_mean" is the average velocity of the device during the test. It is measured in m/s.
Changes in Velocity_mean Index. | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Velocity_mean" is the average velocity of the device during the test. It is measured in m/s.
Changes in the Length_tot Index | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Length_tot" is the global length of the path travelled by the subject during center-out movements. It is measured in meters and it ranges from 0 (no movement) to 2.808 m (patient can fully perform the entire task);
Changes in the Length_tot Index | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Length_tot" is the global length of the path travelled by the subject during center-out movements. It is measured in meters and it ranges from 0 (no movement) to 2.808 m (patient can fully perform the entire task);
Changes in the Score Index. | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Score" is the mean of the ratios between the actual distance covered by the patients and the required distance to be travelled, computed for each required movement; it ranges from 0 (no movement) to 10 (the patient can fully perform the required task). It is a dimensionless index.
Changes in the Score Index. | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Score" is the mean of the ratios between the actual distance covered by the patients and the required distance to be travelled, computed for each required movement; it ranges from 0 (no movement) to 10 (the patient can fully perform the required task). It is a dimensionless index.
Changes in the Work_tan Index. | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Work_tan" is the amount of total work directed towards the target. It is measured in Joules.
Changes in the Work_tan Index. | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinematics of the end-effector of the robot will be acquired during reaching tasks performed by the patient without any assistance from the device. Specifically, "Work_tan" is the amount of total work directed towards the target. It is measured in Joules.
Changes in kinetic parameters: Force (N) towards 8 targets | Before the intervention, after a 3-week robotic rehabilitation intervention
  The kinetics of the end-effector of the robot will be measured by the robot during reaching tasks performed by the patient against the device. The outcome will be the maximum values towards 8 targets.
Changes in kinetic parameters: Force (N) towards 8 targets | Before the intervention, after a 6-week robotic rehabilitation intervention
  The kinetics of the end-effector of the robot will be measured by the robot during reaching tasks performed by the patient against the device. The outcome will be the maximum values towards 8 targets.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Aprile, MD, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Santa Maria della Provvidenza Center, Rome, Italy